CLINICAL TRIAL: NCT06619223
Title: Ankle Arterial Doppler Waveform Assessment For Surveillance Following Lower Limb Revascularisation
Acronym: WAVE
Status: Not yet recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 24SM8819
Record Dates: First submitted 2024-09-20; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; Surveillance; ultrasound
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Ultrasonography, Doppler, Duplex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Duplex Ultrasound — The primary intervention in this study is the use of ankle Doppler waveform assessment for post-revascularisation surveillance in patients with Peripheral Arterial Disease (PAD). This technique utilises continuous-wave Doppler (CWD) and pulsed-wave Doppler (PWD) to assess the blood flow in the key ankle arteries, including the dorsalis pedis artery (DPA) and posterior tibial artery (PTA).

SUMMARY:
The goal of this observational study is to determine the diagnostic performance of serial ankle arterial Doppler waveform assessments in detecting significant arterial restenosis in patients with Peripheral Arterial Disease (PAD) undergoing lower limb revascularization. The main questions it aims to answer are:

Can serial ankle Doppler waveform assessments accurately detect restenosis following revascularization? How cost-effective is this method for long-term patient surveillance? Researchers will compare the results of serial visual Doppler waveform assessments (handheld continuous-wave and pulsed-wave Doppler) with full lower limb arterial duplex ultrasound (DUS) to determine if the Doppler devices provide a comparable diagnostic performance.

Participants will:

Undergo regular pre- and post-revascularization ankle waveform assessments. Participate in follow-up surveillance visits at 3, 6, and 12 months.

DETAILED DESCRIPTION:
This study is a single-centre, prospective observational diagnostic accuracy study designed to evaluate the effectiveness of serial ankle arterial Doppler waveform assessments for post-revascularisation surveillance in patients with Peripheral Arterial Disease (PAD). The study will compare Doppler waveform assessments using both handheld continuous-wave Doppler and pulsed-wave duplex ultrasound (PWD) against a full lower limb duplex ultrasound (DUS), which serves as the reference standard.

Study Procedures:

The study involves a series of non-invasive, repeatable tests that monitor blood flow in the ankle arteries. The following arteries will be examined at the ankle:

Dorsalis pedis artery (DPA) Posterior tibial artery (PTA)

Waveforms are captured and analysed using both auditory and visual outputs from the Doppler devices. Pathological findings, such as monophasic waveforms (indicative of restenosis), will be compared to the normal biphasic or triphasic waveforms.

Index Tests:

Handheld Continuous-Wave Doppler (CWD):

A continuous signal captures real-time blood flow velocity. Visual and audio Doppler signals will be recorded, and waveform morphology will be assessed.

Waveforms will be stored on an external memory device for later analysis.

Pulsed-Wave Doppler (PWD) Duplex Ultrasound:

Provides detailed spectral waveform analysis of ankle vessels using a Doppler angle <60° to assess the velocity and shape of blood flow.

Key parameters such as peak systolic velocity (PSV) will be measured to detect stenosis.

Reference Test:

Full Lower Limb Arterial Duplex Ultrasound (DUS):

Conducted on all patients as part of routine care. Measures Peak Systolic Velocity (PSV) and PSV ratio at areas of suspected stenosis, covering the entire lower limb from the iliac to tibial arteries.

Data Collection:

Data will be collected during pre- and post-revascularisation procedures, and participants will undergo follow-up surveillance at 3, 6, and 12 months. The study will also assess the cost-effectiveness of using ankle Doppler assessments as a substitute for full lower limb DUS, with an evaluation of patient acceptability through Likert scale surveys.

Reliability Measures:

To ensure robustness, inter- and intra-rater reliability will be evaluated through repeated tests by the same and different operators. Machine learning algorithms will also be applied to classify arterial waveforms based on signal processing techniques.

Sample Size and Statistical Analysis:

The study will recruit 121 patients, with each participant undergoing three surveillance visits post-revascularisation. A total of 362 episodes or visits will be analysed. Sensitivity, specificity, and other diagnostic accuracy measures will be calculated, with Cohen's Kappa used to evaluate agreement between the index and reference tests.

The results of this study could provide a cost-effective, patient-friendly alternative for post-revascularisation surveillance, potentially reducing the need for full DUS exams while maintaining diagnostic accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 18 and above) with diagnosed Peripheral Arterial Disease (PAD).
* Patients scheduled for lower limb revascularisation procedures.
* Patients willing and able to provide informed consent.
* Patients who can attend follow-up visits at 3, 6, and 12 months post-revascularisation.

Exclusion Criteria:

* Patients with non-compressible arteries (due to calcification or other reasons).
* Patients who are unable to undergo Doppler assessments for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients with Peripheral Arterial Disease (PAD) undergoing lower limb revascularisation. The participants will be recruited from three hospitals and will include individuals from diverse demographic backgrounds, focusing on those eligible for surgical revascularisation. The study aims to include both male and female patients, with no restrictions based on race or ethnicity.
Sampling Method: Probability Sample
Enrollment: 121 (Estimated)
Dates: Start 2024-10-10 (Estimated); Primary Completion 2025-10-10 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of Ankle Doppler Waveform Assessment for Detecting Arterial Restenosis | 12 months post-revascularisation
  The primary outcome is the diagnostic sensitivity of serial ankle Doppler waveform assessments (using continuous-wave and pulsed-wave Doppler) for detecting significant arterial restenosis in the dorsalis pedis artery and posterior tibial artery. The sensitivity of the Doppler waveform results will be compared against the reference standard of a full lower limb duplex ultrasound (DUS), performed at baseline and during follow-up surveillance visits post-revascularisation.

SECONDARY OUTCOMES:
Specificity and Predictive Values of Ankle Doppler Waveform for Arterial Restenosis | 12 months post-revascularisation
  The secondary outcome measures include the specificity, positive predictive value (PPV), and negative predictive value (NPV) of serial ankle Doppler waveform assessments in detecting significant arterial restenosis in the dorsalis pedis and posterior tibial arteries. The Doppler waveform results will be compared against full lower limb duplex ultrasound (DUS) to assess the accuracy and clinical utility of this non-invasive method.
Cost-Effectiveness of Ankle Doppler Waveform Assessment | 5 years
  This secondary outcome measure evaluates the cost-effectiveness of using serial ankle Doppler waveform assessments compared to full lower limb duplex ultrasound (DUS) for post-revascularisation surveillance. Cost-related data, including the cost of equipment, personnel, and patient time, will be collected and analysed over a 5-year time horizon, alongside quality-adjusted life years (QALYs) and Incremental Cost-Effectiveness Ratios (ICER).

CONTACTS AND LOCATIONS:
Overall Officials: Alun H Davies, Study Chair — Imperial College London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alodayni HM, Smith S, Poushpas S, Swagell K, Mandic D, Johnson NA, Jaffer U, Davies A, Normahani P. Study protocol for a prospective diagnostic accuracy study to assess the feasibility and diagnostic accuracy of serial ankle handheld Doppler waveform assessment (Ankle HHD) for surveillance after lower-limb revascularisation: WAVE study. BMJ Open. 2025 Sep 30;15(9):e107609. doi: 10.1136/bmjopen-2025-107609. PMID 41033760

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT06619223/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-16): https://cdn.clinicaltrials.gov/large-docs/23/NCT06619223/ICF_001.pdf